### Janssen Research & Development

### **Statistical Analysis Plan**

A Randomized, Multicenter, Double-Blind, Parallel, Placebo-Controlled Study of the Effects of Canagliflozin on Renal Endpoints in Adult Subjects With Type 2 Diabetes Mellitus

The CANVAS-R Trial (CANagliflozin cardioVascular Assessment Study-Renal)

Protocol 28431754DIA4003; Phase 4\*\*

JNJ-28431754 (canagliflozin)

\*\*This is a Phase 4 postmarketing study required by the US Food & Drug Administration but may be considered a Phase 3 study in some countries in which canagliflozin has not been approved.

**Status:** Approved

**Date:** 20 March 2017

**Prepared by:** Janssen Research & Development, LLC

**Document No.:** EDMS-ERI-130850882, 2.0

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TABLE | OF CONTENTS | .2 |
|----------|---------------------------------------------------------|----|
| LIST O | F IN-TEXT TABLES | .3 |
| LIST O | F IN-TEXT FIGURES | .3 |
| SUMMA | ARY OF AMENDMENT | .4 |
| ABBRE | VIATIONS | .5 |
| 1. IN | TRODUCTION | .6 |
| 1.1. | Trial Design | .6 |
| 1.2. | Randomization | .8 |
| 1.3. | Trial Objectives | .8 |
| 1.3.1. | Primary Objective | .8 |
| 1.3.2. | Secondary Objectives | |
| 1.3.3. | Exploratory Objectives | |
| 1.4. | Statistical Hypotheses | |
| | <b>,</b> , | |
| | ENERAL ANALYSIS DEFINITIONS | |
| 2.1. | Analysis Populations | |
| 2.2. | Analysis Sets | 10 |
| 2.3. | Data Handling | 10 |
| 2.3.1. | Censoring Rules | 10 |
| 2.3.2. | Handling of Key Milestone Dates | 10 |
| 2.3.3. | Visit Windows | 11 |
| | UBJECT INFORMATION | |
| 3.1. | Baseline Anthropometric and Demographic Characteristics | |
| 3.2. | Baseline Disease Characteristics | |
| 3.3. | Disposition Information | 13 |
| 3.4. | Extent of Exposure and Follow-Up | 13 |
| 3.5. | Prior and Concomitant Medications | 14 |
| | FFICACY | |
| 4.1. | Primary Efficacy Endpoint | |
| 4.1.1. | Definition | |
| 4.1.2. | Analysis Methods | |
| 4.1.3. | Subgroup Analyses | 15 |
| 4.1.4. | Supportive Analyses | 16 |
| 4.1.4.1. | On-Treatment Analysis | 16 |
| 4.1.4.2. | Additional Supportive Analyses | 16 |
| 4.1.4.3. | Assessment of Missing Data | 17 |
| 4.2. | Secondary Efficacy Endpoints | |
| 4.2.1. | Definition | |
| 4.2.2. | Analysis Methods | |
| 4.2.2.1. | | |
| 4.2.2.2. | | |
| 4.3. | Multiplicity Adjustment | |
| 4.4. | Exploratory Efficacy Endpoints | |
| 4.4.1. | Definition | |
| 4.4.2. | Analysis Methods | |
| 4.4.2.1. | · | |
| 4.4.2.1. | | |
| 4.4.2.1. | , | |
| 4.4.Z.I. | 2. Regression of Albuminuria | 22 |

| 4.4.2.1.3. | Urinary ACR | 22 |
|---|---|---|
| 4.4.2.1.4. | Change in eGFR | |
| 4.4.2.1.5. | eGFR Slope | |
| 4.4.2.2. | Changes in HbA <sub>1c</sub> | |
| 4.4.2.3. | AHA Ütilization | |
| 5. SAF | ETY | <mark>23</mark> |
| 5.1. A | djudicated MACE Events | 23 |
| 5.1.1. | Analysis Methods | |
| 5.1.2. | Supplementary Analysis | <mark>24</mark> |
| 5.2. A | dverse Eventsdverse Events | <mark>24</mark> |
| 5.2.1. | Adverse Event Collection | 25 |
| 5.2.2. | Analysis Methods | 25 |
| 5.2.2.1. | General Adverse Events | 26 |
| 5.2.2.2. | Male Mycotic Genital Infections | <mark>27</mark> |
| 5.2.2.3. | Selected Malignancies | 27 |
| 5.2.2.4. | Photosensitivity | 28 |
| 5.2.2.5. | Venous Thromboembolic Events | 28 |
| 5.2.2.6. | Fracture | |
| 5.2.2.7. | Amputation | 29 |
| 5.2.2.8. | Diabetic Ketoacidosis | 30 |
| 5.2.2.9. | Pancreatitis | 30 |
| 5.3. C | linical Laboratory Tests | |
| | ital Signs | |
| | lectrocardiogram | |
| REFERE | NCES | 32 |
| APPEND | X | 33 |
| Appendix | | |
| Appendix | · | |
| Appendix | | |
| Appendix | | |
| LIST OF | FIN-TEXT TABLES | |
| Table 1: | Summary of Analysis Sets | 10 |
| Table 2: | Time Intervals for Analysis (in clinic) Visit Windows | |
| Table 3: | Adverse Events of Interest | |
| Table 6. | Adverse Evente of Interest | 20 |
| LIST OF | F IN-TEXT FIGURES | |
| | | _ |
| Figure 1: | Diagram of Study Design | <u>7</u> |
| Figure 2: | Follow-up of Randomized Subjects with Respect to the GTED | 7<br>21 |
| | | .)4 |

### **SUMMARY OF AMENDMENT**

Relative to the statistical analysis plan (SAP) dated 20 September 2016, the major amendments made in this version are summarized as follows.

| Applicable | |
|---|---|
| Section(s) | Description of Change(s) |
| 2.2 | The On-Study analysis set was added for MACE and replaced the ITT analysis set for several adverse events of interest. The upper bound of the data period for the On-Treatment analysis set was clarified as last dose plus 2 days for laboratory parameters except ACR. |
| 4.1.3 | Additional subgroups were added for the analysis of ACR progression. |
| 4.1.4.2<br>(4.4.1.2) | To be consistent with the protocol, confirmed progression (regression) is now changed to confirmed progression (regression) plus the unconfirmed progression (regression) from the last ACR measures. |
| 4.1.4.3 | Updated the multiple analysis section |
| 4.2.1 | Consistent with the analytic approach described in the Cardiovascular Endpoint adjudication charter, it is clarified that undetermined death is considered as CV death. |
| 4.2.2.1 | Additional subgroups were added for the analysis of secondary efficacy endpoints. |
| 4.4.1 | Clarified that any adjudicated non-CV death event where the adjudication committee assigned a renal proximate cause is considered a renal death. |
| 4.4.2.1.3 | Mixed model of repeated measure (MMRM) will include baseline and visit interaction. |
| 5.1.2 | Added examination of MACE data in the first 60 and 90 days on the top of the first 30 days analysis. |
| 5.2.2.9 | Added a section on the analysis of adjudicated pancreatitis. |
| Appendix 8 | Additional lab analytes were included in the Pre-defined Limit of Change (PDLC) criteria. |

#### **ABBREVIATIONS**

ACR albumin creatinine ratio

AE adverse event

AFT accelerated failure time model AHA antihyperglycemic agent ANCOVA analysis of covariance

BL baseline

BMI body mass index
CI confidence interval
CSR clinical study report
CV cardiovascular

DBP diastolic blood pressure DKA diabetic ketoacidosis

EAC Endpoint Adjudication Committee

eCRF electronic case report form

eGFR estimated glomerular filtration rate FDA Food and Drug Administration

 $\begin{array}{ll} \text{GTED} & \text{Global Trial End Date} \\ \text{HbA}_{1c} & \text{hemoglobin A}_{1c} \end{array}$ 

HDL-C high-density lipoprotein cholesterol

HR hazard ratio

IDMC Independent Data Monitoring Committee

ITT Intent-to-Treat

IWRS Interactive Web Response System LDL-C low-density lipoprotein cholesterol

LLN lower limit of normal

MACE major adverse cardiovascular event

MedDRA Medical Dictionary for Regulatory Activities

MH medical history
MI myocardial infarction
PDLC Pre-defined Limit of Change

PT preferred term

RAAS renin angiotensin aldosterone system

SAE serious adverse event
SAP statistical analysis plan
SBP systolic blood pressure
SC steering committee
SCr serum creatinine
SD standard deviation

SGLT2 sodium- glucose cotransporter 2

SI standard international
SOC system organ class
T2DM type 2 diabetes mellitus
TEAE treatment-emergent AE
ULN upper limit of normal
UTI urinary tract infection

### 1. INTRODUCTION

Canagliflozin (JNJ-28431754) is an inhibitor of the sodium-glucose co-transporter 2 (SGLT2) that has been developed as an oral anti-hyperglycemic agent (AHA) for the treatment of patients with type 2 diabetes mellitus (T2DM). In March 2013, canagliflozin was approved for marketing by the United States (US) Food and Drug Administration (FDA).

Following market authorization, the sponsor is required to demonstrate that the upper bound of the 2-sided 95% confidence interval (CI) of the cardiovascular (CV) risk ratio of test drug to comparator be less than 1.3 in accord with FDA Guidance on assessing CV safety of AHAs. As a result of the discussions with FDA, 28431754DIA4003 (CANVAS-R) was initiated in January 2014. The design and the subject characteristics of CANVAS-R are purposefully similar to 28431754DIA3008 (CANVAS), an ongoing CV outcome study initiated in December 2009.

This SAP stipulates definitions of analysis sets, key derived variables and statistical methods for analysis of efficacy and safety specific for CANVAS-R based on the latest amendment INT-5 (September 2016) of the protocol.

### 1.1. Trial Design

The CANVAS-R study enrolled the first subject in January 2014. The study recruited 5,812 subjects who met all inclusion criteria and none of the exclusion criteria. Subjects were randomly assigned to initial treatment with canagliflozin 100 mg or matching placebo administered once daily (in a 1:1 ratio). The randomization was balanced by using permutated blocks with no stratification factor. After 13 weeks, the dose of canagliflozin (or matching placebo) may be up titrated from 100 mg to 300 mg if the subject requires additional glycemic control, provided the 100 mg dose is well tolerated. The CANVAS and CANVAS-R studies will complete when the last subject randomized has approximately 78 weeks of follow-up or when 688 MACE are accumulated between both studies (estimated to occur between January 2017 and April 2017). The announcement of the GTED will mark the anticipated date on which one of these requirements for ending the study will occur.

Following announcement of the projected GTED, for subjects who remain on double-blind study drug, sites will be required to schedule the End of Treatment (EOT) and the 30-day off-drug follow-up visits as per the Time and Events schedule in the protocol; for subjects who prematurely discontinue study drug, sites will be required to make a final contact (ie, schedule the last follow-up visit) or vital status check as soon as possible after announcement of the GTED. All visits (including the 30-day off-drug follow-up visit) will need to be completed prior to the GTED. A single Steering Committee (SC) and an Independent Data Monitoring Committee (IDMC) have been commissioned for this and the CANVAS study. The SC oversees the study conduct, and the IDMC regularly (and on an ad hoc basis) reviews safety data.

Figure 1 shows an overview of the study design and Figure 2 shows the scheduled follow-up of randomized subjects prior to the GTED.



AHA=antihyperglycemic agent; CV=cardiovascular; HbA<sub>1c</sub>=hemoglobin A<sub>1c</sub>; GTED=global trial end date; R=randomization; T2DM=type 2 diabetes mellitus

Announcement of GTED Subject who continues study drug

Follow-up of Randomized Subjects with Respect to the GTED



Note: Following the announcement of the GTED, investigators are not expected to continue collecting data for purposes of the clinical trial after the 30-day post-treatment contact.

Figure 2:

In this study, duplicate urinary samples will be collected from 2 consecutive days (first morning void urine samples from the visit day and the day prior to the visit). The scheduled albumin creatinine ratio (ACR) measurements will be made on Day 1 (baseline), Week 26, Week 52, Week 78, Week 104, Week 156 and the last on-drug visit.

### 1.2. Randomization

Central randomization was implemented in this study. Subjects were randomly assigned to 1 of 2 treatment groups based on a computer-generated randomization schedule prepared by an external vendor based on the specification tested by the sponsor before the study. The randomization was balanced by using randomly permuted blocks; the randomization did not incorporate any stratification factors.

### 1.3. Trial Objectives

## 1.3.1. Primary Objective

In subjects with T2DM receiving standard of care but with inadequate glycemic control and at elevated risk of CV events, to assess the effect of canagliflozin compared to placebo on progression of albuminuria.

# 1.3.2. Secondary Objectives

In subjects with T2DM receiving standard of care but with inadequate glycemic control and at elevated risk of CV events, to assess the effect of canagliflozin compared to placebo on:

- The composite endpoint of death from CV causes or hospitalization for heart failure;
- Death from CV causes.

### 1.3.3. Exploratory Objectives

In subjects with T2DM receiving standard of care but with inadequate glycemic control and at elevated risk of CV events, to assess the effect of canagliflozin compared to placebo on:

- Regression of albuminuria;
- Change in estimated glomerular filtration rate (eGFR) from baseline to the last off-drug value;
- Urinary albumin/creatinine ratio (ACR);
- The composite of 40% decrease in eGFR, renal death or requirement for renal replacement therapy;
- The composite of doubling of serum creatinine (SCr), renal death or requirement for renal replacement therapy;
- The composite of 40% decrease in eGFR, renal death, requirement for renal replacement therapy or CV death;

- The composite of doubling of SCr, renal death, requirement for renal replacement therapy or CV death;
- The composite of 40% decrease in eGFR, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;
- The composite of doubling of SCr, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;
- Change in eGFR determined from a between-group comparison of the eGFR slopes using all on-drug measurements (ie, off-drug values will not be included) of eGFR made from the first on-drug measurement to the final on-drug measurement;
- Changes in HbA<sub>1c:</sub>
- Utilization of AHA therapy.

### 1.4. Statistical Hypotheses

The hypotheses in CANVAS-R are to support superiority claims of canagliflozin relative to placebo in reducing the following events:

- Progression of albuminuria;
- The composite endpoint of death from CV causes or hospitalization for heart failure;
- Death from CV causes.

For each endpoint, the following statistical hypothesis on the hazard ratio (HR) of canagliflozin over placebo will be tested:

 $H_0$ : The hazard ratio  $\geq 1.0$ , versus  $H_1$ : The hazard ratio  $\leq 1.0$ 

Canagliflozin will be claimed to be superior in the reduction of the target events as compared to placebo if the upper bound of 95% CIs of the hazard ratio is less than 1.0.

#### 2. GENERAL ANALYSIS DEFINITIONS

### 2.1. Analysis Populations

- Randomized subjects—subjects who are randomized via the Interactive Web Response System (IWRS);
- Treated subjects—randomized subjects who received at least one dose of double-blind study medication.

For efficacy analyses and baseline summaries, subjects will be analyzed according to their randomization assignment. For safety analysis (eg, adverse events [AEs]) and summary of exposure, subjects will be analyzed according to the predominant treatment received (defined as the treatment to which the subject was exposed for the greatest duration), in the event that subjects receive a treatment other than the one to which they were randomized. The treatment groups referred in this SAP will be all canagliflozin and placebo.

### 2.2. Analysis Sets

Analysis sets consist of 2 components: 1) analysis population (Section 2.1), which specifies the subjects included in an analysis; 2) data period, defining the time window during which data will be included in the analysis.

Table 1: Summary of Analysis Sets

| Analysis Set | Analysis Population | Data Period |
|---|---|---|
| ITT | Randomized subjects | Day 1 to the last trial contact date (see Section 2.3.2) |
| | | up to the GTED |
| On-Study | Treated subjects | Day 1 to the last trial contact date (see Section 2.3.2) |
| | | up to GTED |
| On-Treatment | Treated subjects | Day 1 to the last dose date (see Section 2.3.2) plus X <sup>a</sup> |
| | _ | days or the last trial contact date, whichever is earlier. |

X is 2 days for laboratory (except ACR) and vital sign measurements, and 30 days for CV and mortality endpoints, and adverse events (AEs).

### 2.3. Data Handling

### 2.3.1. Censoring Rules

For each analysis set, events that occur any time during the data period of the corresponding analysis set (see Table 1) will be considered as eligible events; otherwise subjects not experiencing an event will be censored at the earlier of the last trial contact day or end of the respective data period, if not otherwise specified.

# 2.3.2. Handling of Key Milestone Dates

- Trial reference start date (Day 1): the first double-blind dose date for each subject (First dose date). If missing or incomplete, the first dose date will be imputed as the randomization date.
- Last dose date: the date on which the last dose of double-blind study drug was taken by the subject. If only the day is missing, impute the last day of the month. If the month or the year is missing, impute the date as the date of the scheduled visit subsequent to the last visit when the study drug was dispensed. The imputed last dose date should be no later than the end of treatment visit date or the last trial contact date. In addition, the imputed last dose date should be no earlier than the first dose date. The last dose date is the date of permanent study drug discontinuation regardless of any temporary drug interruption.
- Last trial contact date: the date when the last trial-related procedure is conducted. It is defined as the latest of:
  - The date of last visit (scheduled or unscheduled visit; office or phone visit), or
  - The latest known date of an adverse event (AE) or the study endpoint event status, concomitant medication, vital sign measurements or laboratory results as reported on their respective electronic case report form (eCRF), or
  - The date of alternate contact made (eg, family members, relatives, friends, health care providers, public search) confirming the subject's survival status at the time of the GTED.

For subjects who die during the study, the last trial contact date will be defined as the date of death.

#### 2.3.3. **Visit Windows**

The Time and Events Schedule of the protocol indicates the visit timing and procedures (eg, laboratory, vital signs, and other key safety variables) for each visit; however, the timing of a subject's actual visit may not be exactly as per the protocol indicated target day / visit window. Consequently, for by-visit or over-time summaries, depending on the time period(s) involved in the summaries, the conventions outlined below will be used to allocate the data collected at each actual visit to a planned protocol visit by defining visit windows.

Baseline will be defined as the pre-dose measurement closest to or including Day 1 (prior to dose administration). If the pre-dose measurement on Day 1 is missing, the missing value will be imputed by the latest available measurement prior to Day 1. For serum creatinine, the average of the last 2 pre-dose measurement will be used as baseline.

If a subject has 2 or more actual visits in one analysis visit window, the visit closest to the target day will be used as the study visit for that analysis visit window. However, results from all visits will be included in the safety analyses (eg, pre-defined limits of change analysis) to assure that all results are included. If 2 study visits are the same number of days from the target day within the same visit window, the later visit will be considered the study visit for that target day. Even though all visits will be allocated an analysis visit window, only planned protocol visits for each variable will be included in the by-visit summaries or repeated measure analyses.

Note that the algorithms for calculating visit windows are the same for all the data periods (see Table 1). Table 2 summarizes the analysis visit windows for laboratory, vital signs, and other key safety variables.

| Table 2: | Time Intervals for Analysis (in clinic) Visit Windows | | |
|---|---|---|---|
| | duled Visit Time<br>bel on output) | Time Interval<br>(Day) <sup>a</sup> | Target T<br>Point (D |
| (Ia | Baseline | (Day)<br><1 <sup>b</sup> | 1 01111 (1) |

| Scheduled Visit Time<br>(label on output) | Time Interval (Day) <sup>a</sup> | Target Time Point (Day) |
|---|---|---|
| Baseline | ≤1 <sup>b</sup> | 1 |
| Week 13 | 1° –137 | 92 |
| Week 26 | 138–229 | 183 |
| Week 52 | 230–456 | 365 |
| Week 78 | 457–638 | 547 |
| Week 104 | 639–820 | 729 |
| Week 130 | 821–1002 | 911 |
| Week 156 | 1003–1184 | 1093 |
| Week 182 | 1185–1366 | 1275 |
| Week 208 | 1367–1548 | 1457 |

Relative to the day of the first dose of double-blind study drug.

Up to the first dose of double-blind study drug.

Immediately following the first dose of double-blind study drug. For variables with no time or reference collected at baseline, the first window after baseline starts on Day 2 according to the protocol.

#### 3. SUBJECT INFORMATION

# 3.1. Baseline Anthropometric and Demographic Characteristics

Baseline anthropometric and demographic characteristics will be summarized by treatment group. Descriptive statistics (N, mean, standard deviation [SD], median, and range) will be provided by treatment group for the baseline age and baseline body weight.

Additionally, the number and percentage of subjects in the categories of the following variables at baseline will also be summarized by treatment group:

- Age group:  $<65, \ge 65$  years old;
- Sex: Male, Female;
- Race: White, Black or African American, Asian, Others;
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino, Unknown, Not reported;
- Region: North America, Central/South America, Europe, Rest of the World.

### 3.2. Baseline Disease Characteristics

Descriptive statistics (N, mean, SD, median, and range) will be provided by treatment group and overall for the following baseline continuous variables: duration of diabetes (in years), baseline eGFR, baseline ACR, systolic blood pressure (SBP), weight, body mass index (BMI), HbA<sub>1c</sub>, LDL-C, HDL-C, triglycerides, total cholesterol and LDL-C/HDL-C.

Additionally, the number and percentage of subjects will be summarized by treatment group and overall for the following:

- Baseline BMI categories ( $<30, \ge 30 \text{ kg/m}^2$ );
- Currently daily cigarette smoker: Yes/No;
- Baseline  $HbA_{1c} \ge 8\%$ : Yes/No;
- Duration of T2DM  $\geq$  10 years: Yes/No;
- Baseline systolic blood pressure categories (≤140, >140 mmHg);
- Baseline LDL-C categories (≤70, >70 mg/dL);
- Baseline HDL-C categories (<39, ≥39 mg/dL);
- Baseline eGFR categories (<30, 30 to <60, 60 to <90, ≥90 mL/min/1.73m<sup>2</sup>);
- Baseline albuminuria category:
  - Normoalbuminuria (0 ≤ ACR <30 mg/g); Microalbuminuria (ACR ≥30 mg/g and ≤300 mg/g); Macroalbuminuria (ACR >300 mg/g: ACR >300 mg/g and ≤3000 mg/g, ACR > 3000 mg/g).
- History of hypertension: Yes/No;
- History of CV disease: Yes/No;

- History of coronary artery disease: Yes/No;
- History of cerebrovascular disease: Yes/No;
- History of peripheral vascular disease: Yes/No;
- History of heart failure: Yes/No;
- Microvascular diabetes complications (Any, 1, 2 or 3 of retinopathy, neuropathy [diabetic or automatic neuropathy] and nephropathy)
- History of fracture: Yes/No;

The number and percentage of subjects with a history of medical conditions by system organ class and preferred term (based upon the general medical history eCRF) will be summarized by treatment group and overall.

### 3.3. Disposition Information

Disposition will be summarized for all randomized subjects by treatment group using the categories listed below:

- Screen failure;
- Subjects who are randomized (ITT);
- Subjects who are treated;
- Subjects who completed the study (ie, defined as having been followed until a time point between the notification of the GTED and the GTED, or if the subject had died prior to the GTED);
- Subjects who prematurely discontinued study medication;
- Subjects without final vital status.

The reasons for non-randomization, withdrawal from study (eg, lost to follow-up, consent withdrawal), and discontinuation from study medication will be summarized. The distribution of time to premature discontinuation of study medication will be displayed using a Kaplan-Meier plot, where one minus the survival function will be shown.

Listings will be provided for subjects whose predominant treatment differs from their randomized treatment.

### 3.4. Extent of Exposure and Follow-Up

Total exposure time for each subject is defined as the number of days from Day 1 to the last dose date (inclusive), regardless of any temporary drug interruption(s). Follow-up time is defined as the number of days from Day 1 to the last contact day (inclusive) for each subject. Descriptive statistics (N, mean, SD, median, and range) for total exposure or follow-up time will be presented by treatment group.

The number of subjects with duration in each of the following categories (<13 weeks, 13 to <26 weeks, 26 to <52 weeks, 52 to <104 weeks, 104 to <156 weeks,  $\ge156$  weeks) will also be presented by treatment group as well as overall.

### 3.5. Prior and Concomitant Medications

Concomitant medications of interest is collected on the eCRF at baseline and at each on-drug visit. The number of subjects receiving medication in pre-specified categories, such as insulin, sulphonylurea, metformin, statin, anti-thrombotic, diuretic (loop, and non-loop), renin angiotensin aldosterone system (RAAS) inhibitor, will be presented by treatment group at baseline and during on-drug period. In addition, SGLT2 inhibitor use during the off-drug follow-up period will be summarized by treatment group.

### 4. EFFICACY

The analysis will be performed based on the ITT analysis set, if not otherwise specified.

All statistical tests, except those for the primary and secondary efficacy endpoints, will be considered nominal and reported with a 2-sided 95% confidence level.

Unless otherwise stated, all efficacy analyses and summaries will be performed using the treatment groups assigned by IWRS.

### 4.1. Primary Efficacy Endpoint

Subjects without baseline and/or post-baseline ACR measurements will be excluded from the primary efficacy analysis. Furthermore, subjects with macroalbuminuria at baseline (ACR >300 mg/g) will also be excluded from the analysis.

#### 4.1.1. Definition

The primary efficacy endpoint is the time to the first occurrence of progression of albuminuria.

Urinary albumin creatinine ratio (ACR) is used to assess albuminuria. Subjects will be classified as having normoalbuminuria (ACR <30 mg/g), microalbuminuria (ACR  $\ge$ 30 mg/g and  $\le$ 300 mg/g), or macroalbuminuria (ACR of >300 mg/g]).

Progression is the development of microalbuminuria or macroalbuminuria in a subject with baseline normoalbuminuria or the development of macroalbuminuria in a subject with baseline microalbuminuria, accompanied by an ACR value increase of greater than or equal to 30% from baseline.<sup>3</sup>

If the ACR at a visit meets the definition of progression as described, a confirmatory ACR collection approximately 1 to 2 months later (or sooner under unusual circumstances, eg, subject is stopping study drug) should be done. In cases where a confirmatory sample is not collected within 1 to 2 months, the next available set of ACR measurements can be used for confirmation.

The primary efficacy analysis will be based on results of ACR measurements from a single visit whether confirmed or unconfirmed. The date of the progression/regression event will be defined as the visit date of the first urine sample for the potential progression/regression findings. A sensitivity analysis (see Section 4.1.4.2) will be based on results of ACR measurements from a single visit that were confirmed at a subsequent visit.

### 4.1.2. Analysis Methods

At each visit, the geometric mean of the duplicate measurements will be computed and used for all subsequent analyses unless otherwise specified. For ACR values below the lower quantifiable limit, the lower quantifiable limit itself will be used in the geometric mean calculation.

As the primary analysis for the primary efficacy endpoint, the time from Day 1 to first visit date observing progression (ie, using the visit date of the original sample collection and not using the visit date of the confirmatory sample collection) of albuminuria will be analyzed using a Cox proportional hazards regression model. The response variable in the model is time to progression and the model will include treatment and baseline albuminuria status as the explanatory variables. The hazard ratio of canagliflozin compared to placebo and its 95% CI will be estimated. Canagliflozin will be considered superior to placebo in the reduction of progression if the p-value of the test of significance, ie, the Wald test from the Cox model specified above, is  $\leq 0.05$  in the context of multiplicity adjustment described in Section 4.3.

For ITT analysis, endpoint events that occur during the data period (see Table 1) will be considered as eligible events; otherwise subjects will be censored at the last ACR measurement up to GTED.

# 4.1.3. Subgroup Analyses

The homogeneity of treatment effect on the occurrence of the primary endpoint across subgroups will be examined (at a 2-sided significance level of 0.05) via a test for the treatment by subgroup interaction by adding this term and the subgroup as covariates (treated as class variables) to the primary efficacy analysis (Section 4.1.2) model. Subgroup analysis will be conducted when the total number of events is greater than 10 for two treatment groups (all canagliflozin group and placebo) and at least 1 event in both groups. Factors exhibiting interactions at a significance level of p < 0.05 will be identified as suggesting treatment effect heterogeneity, recognizing the multiplicity in testing multiple subgroups such that one or more p-values < 0.05 may be expected to be observed by chance alone.

If a significant interaction is observed, the Gail-Simon test will be used to further examine the nature of the interaction (qualitative or quantitative).

The hazard ratio of canagliflozin (all canagliflozin group) compared to placebo and its 95% confidence interval will be estimated for each of the following subgroups:

- Age group:  $<65, \ge 65$  years old;
- Sex: Male, Female;

- Race: White, Black or African American, Asian, Other;
- Region: Central/South America, Europe, North America, Rest of the World;
- Baseline BMI categories ( $<30, \ge 30 \text{ kg/m}^2$ );
- Baseline composite blood pressure categories ([SBP<140or DBP<90 mmHg] vs. [SBP ≥ 140 and DBP ≥90 mmHg]);</li>
- Baseline eGFR categories (30 to <60, 60 to <90, ≥90 mL/min/1.73m<sup>2</sup>);
- Baseline HbA<sub>1c</sub> ≥8%: Yes/No;
- Baseline albuminuria: Normoalbuminuria, Microalbuminuria;
- Duration of diabetes  $\geq 10$  years: Yes/No;
- History of CV disease: Yes/No;
- Baseline use of Renin angiotensin aldosterone system (RAAS) inhibitor: Yes/No.

### 4.1.4. Supportive Analyses

If not otherwise specified, the supportive analyses will use the same analysis set as in the primary efficacy analysis.

### 4.1.4.1. On-Treatment Analysis

For On-Treatment analysis, endpoint events that occur within the data period (see Table 1) will be eligible events; otherwise subjects will be censored at the earliest of the last ACR measurement date, last study drug dose date + 30 days, or GTED.

The Cox model for primary analysis (as described in Section 4.1.2) will be repeated using the On-Treatment analysis set.

# 4.1.4.2. Additional Supportive Analyses

Several Cox models analogous to the primary efficacy analysis model will also be performed for exploratory purposes:

- The first Cox proportional hazards model involves the use of confirmed progression, plus the unconfirmed progression from the last ACR values;
- Secondly, there will be an analysis that only excludes subjects with baseline nephrotic range macroalbuminuria (ie, ACR > 3000 mg/g). This analysis will evaluate time to first occurrence of ≥1 step progression in the following categories (ie, baseline normoalbuminuria, baseline microalbuminuria, baseline non-nephrotic range macroalbuminuria).

Additionally, the actual onset time of progression of albuminuria can be determined to occur within an interval from a sequence of examination times (ie, data are interval censored). The accelerated failure time (AFT) model with log normal error structure will be implemented considering interval censoring excluding subjects with baseline macroalbuminuria.<sup>4</sup> The dependent variable in the AFT model is the logarithm of time to progression of albuminuria,

expressed as time intervals. The model will include treatment group and baseline albuminuria status as the explanatory variables.

The cumulative progression rate derived from Kaplan-Meier estimate will be displayed graphically to evaluate the timing of progression and the consistency of the treatment effect over time.

### 4.1.4.3. Assessment of Missing Data

The potential impact of missing data in the interpretation of the primary efficacy analysis will be explored. The primary efficacy endpoint, progression of albuminuria was derived from urinary albumin/creatinine ratio (ACR) laboratory measurements which were generally collected biannually while subjects were on treatment (ie on treatment period) up to the global trial end date (GTED). For subjects who discontinue from treatment early before the development of progression of albuminuria, unobserved data of post-baseline ACR measurements at each scheduled visit up to the GTED will be considered missing and will be imputed. The multiple imputation procedure will apply to ACR data and the time to ACR progession data will then be generated based on the imputed data at the schedule visits.

## Data for model development

Due to the staggered enrollment of the study, for those randomized at a later stage of the enrollment period, pseudo visits up to the max possible visit week prior to GTED, i.e. week 130, will be created according to the protocol schedule. In addition, multiple data points at each visit, e.g. confirmatory samples, will be aggregated using geometric mean according to the variability of ACR data. There is small proportion of subjects (less than 2.5%) with unscheduled visits which will be combined with the closest scheduled visit using the same approach.

### Imputation model

Assuming that after treatment discontinuation, subjects discontinued from the canagliflozin arm will exhibit a response similar to subjects in the placebo arm, the imputation model will be fit using the non-missing data in the placebo group and adjusted for covariates that may be related to the missing data mechanism and the risk of progression based on clinical judgment. The potential covariates include:

- Baseline ACR (continuous);
- Baseline eGFR categories (30 to <60, 60 to <90, ≥90 mL/min/1.73m<sup>2</sup>);
- Baseline blood pressure (SBP<140, DBP<90 mmHg): Yes/No;</li>
- Baseline  $HbA_{1c} \ge 8\%$ : Yes/No;
- Age group:  $<65, \ge 65$  years old;
- Race: White, Other;
- Sex: Male, Female;

In case of convergence issues, the covariates will be removed from the model in the descending order of the list (ie, starting from the bottom of the list).

Due to the highly skewed data of ACR, both baseline and post baseline ACR in the imputation model will be log transformed.

### **Imputation Procedures**

There are about 3% of subjects with intermittent missing in post-baseline ACR data. Those missing data will be imputed with data estimated from all observed data using the Markov Chain Monte Carlo procedure such that the missing data pattern is monotonic.

The post-treatment ACR data increased gradually over time from the end-of-treatment data. Therefore, a "copy control" strategy will be applied and the imputation model will be fit sequentially at each visit using non-missing data in the placebo arm and any preceding visits (O'Kelly and Ratitch 2014, Section 7.4.2)<sup>5</sup>. The estimates of the model parameters are then used to parameterize a Bayesian posterior distribution. At each imputation, missing data in both active and placebo arms will be replaced with predicted values randomly drawn from the distribution. The imputed data will also be applied to the models of subsequent visits. For example, the imputation model at week 26 will be fit using baseline and covariate data (see Section of Imputation Model) and week 26 data of the placebo arm. The ACR data that are missing at week 26 in both active and treatment arms will be imputed in the same way. Similarly, the imputation model for week 52 will utilize observed data of control arm at week 52 and all the preceding data points, whether imputed or observed.

For subjects with missing data, the imputed data up to the earlier of death date or GTED will be combined with observed data. For subjects completing the treatment or developing progression, only data imputed for intermittent missing will be added back to the observed data.

#### Re-construction of time to progression data

The time to progression will be re-defined based on the imputed dataset where subjects with imputed or observed ACR that met the progression criteria will be considered having events at the corresponding visit. Subjects remaining event-free will be censored at the last scheduled visit before death date or GTED, whichever is earlier.

#### **Analysis summary**

The imputed data will be re-analyzed using the same Cox model for the primary analysis (see Section 4.1.2). The imputation process will be repeated 1000 times and the multiple versions of analysis results will be combined into single inferential summary using Rubin's rule.

### 4.2. Secondary Efficacy Endpoints

#### 4.2.1. Definition

There are 2 secondary efficacy endpoints specified in this study:

- The composite endpoint of death from CV causes or hospitalization for heart failure;
- Death from CV causes (CV Death).

Analyses will be using adjudicated events and adjudication of these outcomes by the Endpoint Adjudication Committee (EAC) will be done in a blinded fashion.

### 4.2.2. Analysis Methods

The analyses will be using the ITT analysis set.

### 4.2.2.1. The Composite of CV Death or Hospitalization for Heart Failure

The analysis will be based on time to the first occurrence of the composite event using ITT analysis set. The hazard ratio of canagliflozin compared to placebo and its 95% CI will be estimated using a stratified Cox proportional hazards regression model with treatment as the explanatory variable and history of CV disease (secondary and primary prevention) as the stratification factor. The p-value from the stratified log rank test for the treatment effect will also be reported.

The subgroup analysis will be conducted using the same approaches described in Section 4.1.3 and the following subgroups:

- Age group:  $<65, \ge 65$  years old;
- Sex: Male, Female;
- Race: White, Black or African American, Asian, Other;
- Region: Central/South America, Europe, North America, Rest of the World;
- Baseline BMI categories ( $<30, \ge 30 \text{ kg/m}^2$ );
- Baseline composite blood pressure categories ([SBP <140 or DBP <90 mmHg] vs. [SBP ≥140 and DBP ≥90 mmHg]);
- Baseline eGFR categories (30 to <60, 60 to <90, ≥90 mL/min/1.73m<sup>2</sup>);
- Baseline  $HbA_{1c} \ge 8\%$ : Yes/No;
- Duration of diabetes ≥ 10 years: Yes/No;
- History of CV disease: Yes/No;
- History of peripheral vascular disease: Yes/No;

19

<sup>&</sup>lt;sup>a</sup> Undetermined death is considered CV death.

- History of amputation: Yes/No;
- Baseline use of statin;
- Baseline use of anti-thrombotics;
- Baseline use of RAAS inhibitor;
- Baseline use of Beta blocker;
- Baseline use of insulin;
- Baseline use of diuretics.

### 4.2.2.2. CV Death

The analysis will be based on time to the first occurrence of CV death using ITT analysis set. The hazard ratio of canagliflozin compared to placebo and its 95% CI will be estimated using a stratified Cox proportional hazards regression model with treatment as the explanatory variable and history of CV disease (secondary and primary prevention) as the stratification factor. The p-value from the stratified log rank test for the treatment effect will also be reported.

Subgroup analyses will be performed using the same subgroups and the analysis methods described in Section 4.2.2.1.

### 4.3. Multiplicity Adjustment

Per the SAP of the integrated summary of CANVAS and CANVAS-R studies, only one alpha family is proposed for the testing of the multiple hypotheses based on the integrated data and the CANVAS-R data. The Type I error for these tests will be strictly controlled via a gatekeeping procedure. If the MACE and the mortality endpoints in the integrated analysis succeed in rejecting the null hypotheses, all of the alpha for testing (ie, 5%) will pass to the CANVAS-R for testing of the primary and the secondary hypotheses of the study. Tests for CANVAS-R hypotheses will proceed sequentially conditional on the statistical significance of the hypothesis tests in the integrated summary at the 5% significant level.

Figure 3: Hypothesis Testing Sequence



### 4.4. Exploratory Efficacy Endpoints

### 4.4.1. Definition

The following exploratory endpoints will be analyzed:

- Time to the first occurrence of composite endpoint of 40% decrease in eGFR, renal death<sup>a</sup> or requirement for renal replacement therapy;
- Time to the first occurrence of composite endpoint of doubling of SCr, renal death or requirement for renal replacement therapy;
- Time to the first occurrence of composite endpoint of 40% decrease in eGFR, renal death, requirement for renal replacement therapy or CV death;
- Time to the first occurrence of composite endpoint of doubling of SCr, renal death, requirement for renal replacement therapy or CV death;
- Time to the first occurrence of composite endpoint of 40% decrease in eGFR, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;
- Time to the first occurrence of composite endpoint of doubling of SCr, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;
- Regression of albuminuria;

Regression of albuminuria is the development of normoalbuminuria in a subject with baseline microalbuminuria or macroalbuminuria or the development of microalbuminuria in a subject with baseline macroalbuminuria, accompanied by a decrease in the ACR value of greater than or equal to 30% from baseline. If the ACR at a visit meets the definition of potential regression described above, a confirmatory ACR collection approximately 1 to 2 months later

<sup>&</sup>lt;sup>a</sup> Non-CV death with a renal proximate cause is considered as renal death.

(or sooner under unusual circumstances, eg, subject is stopping study drug), should be done. In cases where a confirmatory sample is not collected within 1 to 2 months, the next available set of ACR measurements can be used for confirmation.

- Change in urinary ACR over time;
- Change in eGFR from baseline to the last off-drug measurement;
- Estimated eGFR slopes using all on-drug measurements;
- Changes in HbA<sub>1c</sub>.
- AHA utilization

# 4.4.2. Analysis Methods

### 4.4.2.1. Renal Endpoints

### 4.4.2.1.1. Composite Endpoints

The components of the renal composite endpoints, such as requirement for renal replacement therapy and doubling of serum creatinine, identified by the investigator or the sponsor for meeting the criteria pre-specified in the charter will be sent to the independent EAC.

The time to the first occurrence of each of the renal composite endpoints (see Section 4.4.1) will be analyzed in the ITT analysis set using a Cox proportional hazards model with treatment and baseline eGFR ( $< 60, \ge 60 \text{ mL/min/1.73m}^2$ ) as the explanatory variables. The hazard ratio of canagliflozin compared to placebo and its 95% confidence interval will be estimated from the model.

### 4.4.2.1.2. Regression of Albuminuria

Regression of albuminuria will be analyzed in a similar fashion in modeling and censoring rule as the analysis for progression of albuminuria. The analysis will be using the ITT analysis set based on ACR measurements from a single visit whether confirmed or unconfirmed. Subjects with normal albuminuria at baseline will be excluded. The hazard ratio of canagliflozin compared to placebo and its 95% confidence interval will be estimated from the model. Additionally, analyses based on confirmed regression plus unconfirmed regression from the last ACR values will be performed in a similar fashion using ITT analysis set.

### 4.4.2.1.3. Urinary ACR

Post-baseline ACR will be analyzed using mixed effect model repeat measurement (MMRM) and the ITT analysis set.

Since the distribution of ACR is highly skewed, the log transformed ACR values of all the post-baseline and scheduled visits will be modeled, using a linear mixed effects model. The linear mixed effects model will be fit to the logarithm of ACR as a dependent variable, including treatment, logarithm of baseline ACR value, visit, treatment by visit interaction, and logarithm of baseline ACR value by visit interaction as fixed effects. The percentage of treatment difference,

ie, treatment difference in mean ACR relative to placebo, can be calculated by taking the antilogarithm of the estimated coefficient for the treatment group and subtracting 1. The ratio of mean ACR in treatment compared to placebo and its 95% CI will be presented. An unstructured covariance will be used to model the within subject errors.

# 4.4.2.1.4. Change in eGFR

For change in eGFR from baseline to the last off-drug measurement will be analyzed in the ITT analysis set using an analysis of covariance (ANCOVA) model with treatment and the baseline eGFR value as covariates. The treatment difference of canagliflozin compared to placebo in the least-squares means and associated 95% CI will be estimated from the model.

# 4.4.2.1.5. eGFR Slope

The time slope of eGFR will be analyzed in the On-Treatment analysis set using a linear mixed effects model with eGFR as a dependent variable and treatment, baseline eGFR value, time (as a continuous variable), and treatment by time interaction as fixed effects and intercept and time as random effects. The parameter of interest is the coefficient for treatment by time interaction term, which measures the slope difference between canagliflozin and placebo over time.

# 4.4.2.2. Changes in HbA<sub>1c</sub>

Change in HbA<sub>1c</sub> from baseline will be analyzed using MMRM and the ITT analysis set. The effect of canagliflozin relative to placebo on the changes in HbA<sub>1c</sub> from baseline over time will be assessed using MMRM. The analysis will include the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline and baseline-by-visit interaction. An unstructured covariance will be used to model the within subject errors.

#### 4.4.2.3. AHA Utilization

Summary of AHA utilization is described under Section 3.5.

### 5. SAFETY

The safety analysis will be mainly based on the On-Treatment analysis set unless otherwise specified.

There will be no imputation of missing values for clinical laboratory test results, vital sign measurements in the safety analyses.

# 5.1. Adjudicated MACE Events

The MACE is the composite of CV outcomes including CV death, non-fatal MI<sup>a</sup>, or non-fatal stroke. Adjudication of these outcomes by the EAC has been done in a blinded fashion.

<sup>&</sup>lt;sup>a</sup> Silent MIs are excluded from the analysis.

### 5.1.1. Analysis Methods

The analysis will be based on the time to first occurrence of MACE using the ITT analysis set. The HR of all canagliflozin compared to placebo and its 95% CI will be estimated using a stratified Cox proportional hazards regression model with treatment (all canagliflozin and placebo) as the explanatory variable, and prior CV disease subgroup (secondary prevention and primary prevention) as the stratification factors. P-value of stratified log rank test for treatment effect will also be reported for the primary analysis.

### 5.1.2. Supplementary Analysis

A prior post-hoc analysis performed by the FDA of the MACE-plus events occurring during the first 30 days post-randomization in CANVAS showed an imbalance in favor of placebo. In the PMR, FDA requested that the pattern of MACE events occurring in the first 30 days post randomization in CANVAS-R be explored. Additional examination of the MACE events in the first 60 and 90 days using the ITT analysis set will be made.

An excess of volume depletion AEs in the canagliflozin groups could provide a possible biologic basis for an imbalance in MACE events between canagliflozin and control. In the CANVAS study, the Kaplan-Meier (KM) time-to-event analysis comparing canagliflozin and placebo showed that the greatest separation in the curves for volume depletion AEs occurred during the first 90 days post-randomization.

To assess the potential association between MACE events and volume depletion AEs and fulfill the PMR request, hazard ratio will be estimated using the same stratified Cox model as in the main analysis (see Section 5.1.1) for events occurring within the first 30 days, and within the first 90 days post-randomization. In addition, Kaplan-Meier plots including data within first 30 days and first 90 days will be presented.

Additionally, time to the first occurrence of each component of MACE as well as fatal/non-fatal MI and fatal/non-fatal stroke will be analyzed using the same Cox model described in Section 5.1.1.

### 5.2. Adverse Events

Adverse events (AEs) will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) at the time of database lock.

A treatment-emergent AE (TEAE) is defined as an AE with an onset after the initiation of double-blind study drug and before the last study medication date plus 30 days. AEs with a start date prior to initiation of double-blind study drug which are subsequently reported to have either an increase in intensity or change in attribution in relationship to study drug (ie, attribution to possible, probably, very likely) after the initiation of double-blind study drug will also be considered as TEAEs.

#### 5.2.1. Adverse Event Collection

The AE collection in CANVAS-R is streamlined to include serious adverse events (SAEs), AEs that lead to study drug discontinuation, and all AEs (serious and non-serious) for selected AEs of interest (Table 3, Section B).

For selected AEs of interest, additional data will be collected on supplementary CRF pages mainly for the purposes of narrative description of certain events. Table 3 lists the AEs of interest.

#### **Table 3:** Adverse Events of Interest

# Section A: For the AEs listed below, only serious AEs or AEs that led to drug discontinuation were collected:

Osmotic diuresis

Volume depletion

Hypoglycemia

Urinary tract infection (UTI)

Female mycotic genital infection

Severe hypersensitivity /cutaneous reactions

**Pancreatitis** 

Hepatic injury

Renal related AEs (including Nephrotoxicity/ acute kidney injury)

# Section B: The AEs listed below were collected regardless of whether they were serious and/or led to study drug discontinuation for the study:

Male mycotic genital infection (balanitis, phimosis, events leading to circumcision)

Malignancy

Renal cell cancer

Bladder cancer

Pheochromocytoma

Levdig cell tumors

Breast cancer

Photosensitivity

Venous thromboembolic events (VTE)

Amputation

Fracture

Diabetic Ketoacidosis

The AEs listed above will be identified using a MedDRA preferred term list (Appendix 1.3).

# 5.2.2. Analysis Methods

The study duration of CANVAS-R is long relative to the rest of the canagliflozin Phase 3 program. Accordingly, the incidences of AEs (ie, proportion of subjects reporting the AEs) derived from the study are not comparable to the incidences generated in the Phase 3 program. Therefore, the exposure-adjusted incidence rate will be reported in addition to the incidence. The rate is calculated as the total number of subjects with the AE divided by the On-treatment exposure in subject-years. For some particular AEs such as malignancy where the off-drug follow

up is included, the follow-up-adjusted incidence rate will be estimated. The rate is calculated as the total number of subjects with the AEs divided by the total follow-up time in subject-years.

For general AEs and selected AEs of interest that are not routinely collected in CANVAS-R (refer to Section A of Table 3), the main interest will be the serious AEs and the AEs leading to discontinuation of study medication.

#### 5.2.2.1. General Adverse Events

An overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- Serious AEs;
- Deaths;
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

SAEs by system organ class and preferred term will be summarized by treatment group using the On-Treatment analysis set. The same summary will be provided for AE leading to discontinuation of study medication using the On-Treatment analysis set.

The incidence of all SAEs (by preferred term, grouped by SOC, and presented by treatment group) will also be summarized by the relationship to study drug, by the action taken regarding the study drug, as well as by the outcome. The relationship to study drug will be presented by 2 categories: related (which includes possibly related, probably related and very likely related, as reported by the investigator) and not related (which includes not related and doubtfully related, as reported by the investigator).

For reference, as a screening tool, the 95% CIs for incidence difference between treatment groups will be calculated for the AEs which are reported in at least 4 or more subjects in any treatment group. Four (rule-of-4) was chosen based on the recommendation from the Safety, Planning, Evaluation, and Reporting Team (SPERT). The exclusion of "0" from the 95% CI for the between-group difference in incidence for a particular AE does not necessarily imply that the difference is due to drug. The intent of providing the 95% CIs is as a filter to identify AEs that require additional assessment. AEs identified by the above screening procedure will be presented and may be subject to further evaluation.

Listings will also be provided for deaths, SAEs, and AEs leading to study drug discontinuation.

For AEs of interest in Section A of Table 3, a summary similar to the analysis of general AEs will be provided. The AEs will be identified using the MedDRA preferred terms listed in Appendix 1.3.

### **5.2.2.2.** Male Mycotic Genital Infections

Balanitis and phimosis AEs will be identified using the MedDRA preferred terms listed in Appendix 1.3, and the analyses will be based on the On-Treatment analysis set.

An overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- All AEs;
- Serious AEs;
- AEs considered drug-related (investigator assessment of possible, probable or very likely);
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

AEs by preferred term will be summarized by treatment group. A Kaplan-Meier plot for the time to first occurrence of balanitis will be provided by treatment group.

In addition, circumcision events will be identified using the sponsor's pharmacovigilance database and summarized by treatment group.

# 5.2.2.3. Selected Malignancies

The selected malignancies of interest are renal cell cancer, bladder cancer, testicular cancer (Leydig cell tumors), pheochromocytomas, and breast cancer. Selected malignancy AEs will be identified using the MedDRA Preferred terms listed in Appendix 1.3, and the analyses will be based on the On-Study analysis set.

For each selected malignancy of interest, an overview summary table with the incidence and the follow-up-adjusted incidence will be provided for:

- All AEs;
- Serious AEs;
- AEs considered drug-related (investigator assessment of possible, probable or very likely);
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication:
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

The preferred terms associated with each selected malignancy type will be summarized by treatment.

A summary of all malignancy events as reported in the malignancy supplementary page will be reported by treatment and primary site. For breast, bladder, or renal cancers, the risk factors for each cancer type captured in the supplementary page will be summarized by treatment.

# 5.2.2.4. Photosensitivity

Photosensitivity AE will be identified using the MedDRA preferred terms listed in Appendix 1.3, and the analyses will be based on the On-Treatment analysis set.

An overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- All AEs;
- Serious AEs;
- AEs considered drug-related (investigator assessment of possible, probable or very likely);
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

AEs by preferred term will be summarized by treatment group.

#### 5.2.2.5. Venous Thromboembolic Events

Venous thromboembolic (VTE) events will be identified using the MedDRA preferred terms listed in Appendix 1.3.

An overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- All AEs;
- Serious AEs:
- AEs considered drug-related (investigator assessment of possible, probable or very likely);
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

AEs by preferred term will be summarized by treatment group.

#### 5.2.2.6. Fracture

Fracture events identified by the investigator or the sponsor for meeting the criteria pre-specified in the charter will be sent to the independent Fracture Adjudication Committee to confirm that

events were fractures and to determine fracture location (anatomic region) and type (low trauma or not). The main analyses of the adjudicated low trauma fracture AEs will be based on the On-Study analysis set.

An overview summary table with the incidence and the follow-up-adjusted incidence will be provided for:

- Adjudicated fractures;
- Adjudicated fractures considered serious (investigator assessment);
- Adjudicated fractures considered drug-related (investigator assessment of possible, probable or very likely);
- Adjudicated fractures leading to discontinuation of study medication;
- Adjudicated fractures considered serious and drug-related (investigator assessment);
- Adjudicated fractures considered drug-related (investigator assessment) and leading to discontinuation of study medication.

A summary of adjudicated fracture stratified by anatomical region by treatment will be provided. The incidence as well as the incidence rate will be presented.

Adjudicated AEs associated with fall will be summarized by treatment group.

A Kaplan-Meier plot for the time to the first occurrence of adjudicated fracture event will be provided by treatment group. The hazard ratio between canagliflozin (all canagliflozin) compared to placebo and its 95% confidence interval will be estimated from a Cox proportion hazards model with treatment as the explanatory variable.

A summary of all adjudicated fractures by anatomic location will be provided. The hazard ratio and its 95% CI as well as a Kaplan-Meier plot for the first occurrence of all adjudicated fractures will be provided using the same analysis as the adjudicated low trauma fractures.

## 5.2.2.7. Amputation

The main analysis of lower extremity amputations as documented in the dedicated case report form page will be based on the On-Study analysis set. An overview summary table with the incidence and the follow-up-adjusted incidence will be generated for:

- All lower limb amputations;
- Traumatic lower limb amputation;
- Atraumatic lower limb amputation.

Summary of anatomical region (toe, ankle, trans-metatarsal, below knee, above knee) of lower extremity atraumatic amputations will be reported by treatment group.

For atraumatic lower limb amputation, a Kaplan-Meier plot for the time to the first occurrence of event will be provided by treatment group.

For the post-treatment AEs that may be associated with amputation, groupings of selected MedDRA preferred terms used to identify events to be included in each of the following SOC categories are presented in Appendix 1.4:

- Infections and Infestations;
- Vascular disorders;
- Nervous System disorders;
- Skin and subcutaneous tissue disorders;
- Osteomyelitis.

The selected preferred terms in infections and infestation are further split into "Reversible Infection" and "Irreversible Infections". In addition, the preferred terms grouped under the MedDRA high level term of "skin and subcutaneous tissue ulcerations" are also of interest.

For each AE group listed above, the incidence of the respective preferred terms will be summarized by treatment group.

### 5.2.2.8. Diabetic Ketoacidosis

Diabetic ketoacidosis (DKA) and related AEs will be identified using the list of MedDRA terms in Appendix 1.3. Adverse events identified by the investigator or the sponsor for meeting the criteria pre-specified in the charter will be sent to the independent DKA Adjudication Committee. The main analysis of the DKA events will be based on adjudicated events of DKA in the On-Study analysis set. Events occurring at any time post-randomization, regardless of the timing of the last dose of study medication, will be included. For the adjudicated DKA events, a table will summarize the incidence and the follow-up-adjusted incidence rate.

A listing of all DKA and related events identified by the sponsor's medical monitoring team and the subset of these events that went for adjudication will be provided.

#### 5.2.2.9. Pancreatitis

Pancreatitis and related AEs identified by the sponsor using the list of MedDRA terms prespecified in the charter will be sent to the independent Pancreatitis Adjudication Committee. The main analysis of events will be based on adjudicated, confirmed events in the On-Treatment analysis set. Analysis based on events occurring at any time post-randomization, regardless of the timing of the last dose of study medication, will be performed. The incidence rate and proportion of adjudicated pancreatitis events by severity will be summarized. The total number of subjects with an event not confirmed by the Pancreatitis Adjudication Committee will also be summarized.

# 5.3. Clinical Laboratory Tests

A list of clinical laboratory assessments made during the study is provided in Appendix 1.1. The percentage of subjects with specific treatment-emergent laboratory values meeting pre-defined limit of change (PDLC) criteria listed in Appendix 1.2 will be summarized. The 95% CI for the percentage difference between canagliflozin compared to placebo group will be provided for each

PDLC criterion which have at least 4 or more subjects in any treatment group. A corresponding listing will also be provided. As described above, PDLC values will be presented based on measurements on study drug and up to a maximum of 2 days after the last dose of study drug, as well as all measurements regardless of the time of the last dose of double-blind study drug. Summaries based on both standard units (SI) and conventional units will be provided.

# 5.4. Vital Signs

A treatment-emergent vital sign abnormality is defined as a change from baseline and subsequent post-baseline value that satisfies the PDLC criteria in Appendix 1.2. For each vital sign parameter, the proportion of subjects with a treatment-emergent abnormality will be tabulated by treatment group. PDLC values will be presented based on measurements up to a maximum of 2 days after the last dose of study medication.

The blood pressure measurements will be based on the average of the consecutive sitting blood pressure readings that were to be collected at each visit.

# 5.5. Electrocardiogram

Electrocardiogram was not be collected in this study.

### **REFERENCES**

- 1. FDA Guidance for Industry: Diabetes Mellitus Evaluating Cardiovascular Risk in New Anti-diabetic Therapies to Treat Type 2 Diabetes, December 2008.
- 2. KDOQI 2007. National Kidney Foundation Kidney Disease Outcomes Quality Initiative (KDOQI). *Amer J of Kidney Diseases* 2007;49(2, Suppl 2):S1-S180.
- 3. Parving HH, Lehnert H, Bröchner-Mortensen J, Gomis R, Andersen S, Arner P; Irbesartan in Patients with Type 2 Diabetes and Microalbuminuria Study Group.N Engl J Med. 2001 Sep 20;345(12):870-8.
- 4. Ruggenenti P, Fassi A, Ilieva AP, Bruno S, Iliev IP, Brusegan Bergamo Nephrologic Diabetes Complications Trial (BENEDICT) Investigators; Preventing microalbuminuria in type 2 diabetes. *N Engl J Med* 2004; 351:1941–1951.
- 5. O'Kelly M (2014), Ratitch B. Overview of the Imputation Methods. In: Clinical Trials with Missing Data. New York: John Wiley & Sons; 2014.
- 6. Crowe BJ, Xia HA, Berlin JA, et al. Recommendations for safety planning, data collection, evaluation and reporting during drug, biologic and vaccine development: a report of the safety planning, evaluation, and reporting team. *Clin Trials*. 2009;6:430-440.

#### **APPENDIX**

#### **Appendix 1.1: Clinical Laboratory Tests**

The clinical laboratory tests include following panels and assessments:

- Hematology panel
  - o hemoglobin
  - o platelet count
  - o hematocrit
  - o red blood cell (RBC) count
  - o white blood cell (WBC) count with differential
- Serum chemistry panel

o sodium alkaline phosphatase o potassium creatine phosphokinase (CPK) lactic acid dehydrogenase (LDH) o chloride bicarbonate o uric acid o BUN o calcium o creatinine o phosphate o aspartate aminotransferase (AST) o albumin o alanine aminotransferase (ALT) o total protein o gamma-glutamyltransferase (GGT) o magnesium o total bilirubin

- Fasting serum lipid profile (triglycerides, LDL-C, HDL-C, total cholesterol).
- HbA<sub>1c</sub>
- Urinalysis (dipstick analysis; from spot urine collection in the clinic on Day 1; performed at central laboratory; microscopic analysis is not required). Urine glucose will not be measured by the central laboratory
  - o specific gravity ketones
  - pH bilirubin/urobilinogen
  - o protein nitrite
  - blood leukocyte esterase
- Central laboratory will report the estimated glomerular filtration rate (eGFR) according to the Modification of Diet in Renal Disease Study (MDRD) equation (Levey 2006) at study visits when serum creatinine is measured. The 4-variable MDRD eGFR includes serum creatinine, age, race, and sex according to the equation below:

For creatinine in mg/dL:

eGFR (mL/min/1.73 m<sup>2</sup>) = 175 x (serum creatinine)  $^{-1.154}$  x (age)  $^{-0.203}$  x (0.742 if female) x (1.21 if black)

For creatinine in µmol/L:

eGFR (mL/min/1.73m<sup>2</sup>) = 175 x (serum creatinine x 0.0113)  $^{-1.154}$  x (age)  $^{-0.203}$  x (0.742 if female) x (1.21 if black)

# Appendix 1.2: Criteria for Pre-defined Limit of Change (PDLC) and Abnormal Values

| Laboratory Test | Parameter for ANY value and LAST value |
|---|---|
| CHEMISTRY | |
| Albumin | Composite: <lln and="">25% decrease from BL</lln> |
| | Absolute Value: >3X ULN |
| ALT | Absolute Value: >5X ULN |
| | Absolute Value: >8X ULN |
| | Absolute Value: >3X ULN |
| AST | Absolute Value: >5X ULN |
| | Absolute Value: >8X ULN |
| | Composite: ALT >3X ULN and Tbili >2X ULN [with the Tbili elevation >2 X |
| ALT >3X ULN and Tbili >2X ULN | ULN within 30 days of the ALT elevation >3x ULN] |
| | Composite: AST >3X ULN and Tbili >2X ULN [with the Tbili elevation >2 X |
| AST >3X ULN and Tbili >2X ULN | ULN within 30 days of the AST elevation >3x ULN] |
| | Composite: >ULN and > 25% increase from BL |
| Bilirubin | Absolute Value: >2XULN |
| Bicarbonate | Absolute Value: <16 mEq/L |
| Calcium | Composite: >ULN and > 10 % increase from BL |
| Creatinine Kinase | Absolute Value: >1000U/L |
| | Composite: < 80 and decrease>30% from BL |
| eGFR | Change: decrease>50% from BL |
| | Composite: <lln and="">25% decrease from BL</lln> |
| Magnesium | Composite: >ULN and >25% increase from BL |
| Phosphorus | Composite: >ULN and >25% increase from BL |
| | Composite: <lln and="">15% decrease from BL</lln> |
| Potassium | Composite: >ULN and >15% increase from BL |
| | Absolute Value: ≥ 6.5 mEq/L |
| | Composite: <lln and="" decrease="">5 mEq/L or more from BL</lln> |
| Sodium | Composite: >ULN and increase>5 mEq/L or more from BL |
| Uric Acid | Composite: <lln and="">25% decrease from BL</lln> |
| HEMATOLOGY | |
| | Change: ≥ 2 g/dl decrease from BL |
| Hemoglobin | Change: ≥ 2 g/dL increase from BL |
| | Composite: <lln and="" decrease="">25% from BL</lln> |
| Platelets | Composite: >ULN and increase >25% from BL |
| | Composite: < LLN and >25% decrease from BL |
| White Blood Count | Composite: > ULN and >50 % increase from BL |
| VITAL SIGNS | |
| | Absolute Value: ≤50 beats per minute |
| Pulse | Absolute Value: ≥100 beats per minute |
| | Composite: ≥ 20 mm Hg decrease from BL and ≤90 mm Hg |
| Systolic Blood Pressure | Composite: ≥ 20 mm Hg increase from BL and ≥ 160 mm Hg |
| | Composite: ≥ 15 mm Hg decrease from BL and ≤ 50 mm Hg |
| Diastolic Blood Pressure | Composite: ≥ 15 mm Hg increase from BL and ≥ 100 mm Hg |

# Appendix 1.3: List of Preferred Terms for Selected AEs of Interest

| | Female Mycotic Genital | |
|---|---|---|
| Diabetic ketoacidosis | Infections | Fracture |
| Acidosis | Genital candidiasis | Acetabulum fracture |
| Acidosis aggravated | Genital infection | Ankle fracture |
| Acidosis diabetic | Genital infection female | Atypical femur fracture |
| Acidosis metabolic | Genital infection fungal | Atypical fracture |
| Acidosis NOS | Urogenital infection fungal | Avulsion fracture |
| Acute acidosis | Vaginal infection | Bone fragmentation |
| Anion gap acidosis | Vaginal inflammation | Cervical vertebral fracture |
| Blood ketone body | Vulvitis | Chance fracture |
| Blood ketone body increased | Vulvovaginal candidiasis<br>Vulvovaginal mycotic | Clavicle fracture |
| Blood ketone body present | infection | Closed fracture manipulation |
| Diabetes mellitus with ketoacidosis | Vulvovaginitis | Comminuted fracture |
| Diabetes with hyperosmolarity | | Complicated fracture |
| Diabetes with ketoacidosis | | Compression fracture |
| Diabetic acidosis | | Craniofacial fracture |
| Diabetic hyperglycemic coma | | Elevation skull fracture |
| Diabetic hyperosmolar coma | | Epiphyseal fracture |
| Diabetic ketoacidosis | | External fixation of fracture |
| Diabetic ketoacidotic hyperglycemic | | |
| coma | | Facial bones fracture |
| Diabetic metabolic decompensation | | Femoral neck fracture |
| High anion gap metabolic acidosis | | Femur fracture |
| Hyperglycemic seizure | | Fibula fracture |
| Hyperosmolar hyperglycemic state | | Foot fracture |
| Hyperosmolar state | | Forearm fracture |
| Ketoacidosis | | Fracture |
| Ketonuria | | Fracture debridement |
| Ketosis | | Fracture delayed union |
| Metabolic acidosis | | Fracture displacement |
| Metabolic acidosis exacerbated | | Fracture malunion |
| Metabolic acidosis NOS exacerbated | | Fracture nonunion |
| Metabolic acidosis not otherwise | | Frankling main |
| specified (NOS) | | Fracture pain |
| Metabolic acidosis worsened Type I diabetes mellitus with | | Fracture reduction |
| ketoacidosis | | Fracture treatment |
| Type II diabetes mellitus with | | |
| ketoacidosis | | Fractured coccyx |
| | | Fractured ischium |
| | | Fractured maxilla elevation |
| | | Fractured sacrum |
| | | Fractured skull depressed |
| | | Fractured zygomatic arch elevation |
| | | Greenstick fracture |
| | | Hand fracture |
| | | Hip fracture |
| | | Humerus fracture |
| | | Ilium fracture |
| | | Impacted fracture |
| | | Internal fixation of fracture |
| | | Jaw fracture |
| | | Limb crushing injury |
| | | Limb fracture |

| | Female Mycotic Genital | |
|---|---|---|
| Diabetic ketoacidosis | Infections | Fracture |
| | | Loss of anatomical alignment after |
| | | fracture reduction |
| | | Lower limb fracture |
| | | Lumbar vertebral fracture |
| | | Multiple fractures |
| | | Open fracture |
| | | Open reduction of fracture |
| | | Open reduction of spinal fracture |
| | | Osteochondral fracture |
| | | Osteoporotic fracture |
| | | Patella fracture |
| | | Pathological fracture |
| | | Pelvic fracture |
| | | Periprosthetic fracture |
| | | Pubis fracture |
| | | Radius fracture |
| | | Rib fracture |
| | | Sacroiliac fracture |
| | | Scapula fracture |
| | | Skull fracture |
| | | Skull fractured base |
| | | Spinal compression fracture |
| | | Spinal fracture |
| | | Spinal fusion fracture |
| | | Sternal fracture |
| | | Stress fracture |
| | | Thoracic vertebral fracture |
| | | Tibia fracture |
| | | Torus fracture |
| | | Traumatic fracture |
| | | Ulna fracture |
| | | Upper limb fracture |
| | | Wrist fracture |

| Hepatic Injury | Hypoglycaemia | Male Mycotic Genital Infections |
|---|---|---|
| Acute graft versus host disease in liver | Hypoglycaemia | Balanitis |
| Acute hepatic failure | Hypoglycaemic coma | Balanitis candida |
| Acute yellow liver atrophy | Hypoglycaemic seizure | Balanoposthitis |
| Allergic hepatitis | | Balanoposthitis infective |
| Ammonia increased | | Erosive balanitis |
| Ascites | | Gangrenous balanitis |
| Asterixis | | Genital candidiasis |
| Autoimmune hepatitis | | Genital infection |
| Bacterascites | | Genital infection fungal |
| Biliary ascites | | Genital infection male |
| Biliary cirrhosis | | Penile infection |
| Biliary cirrhosis primary | | Posthitis |
| Biliary fibrosis | | |
| Bilirubin excretion disorder | | |
| Biopsy liver abnormal | | |
| Child-Pugh-Turcotte score increased | | |
| Cholaemia | | |
| Cholestasis | | |
| Cholestatic liver injury | | |

#### **Hepatic Injury**

#### Hypoglycaemia

#### **Male Mycotic Genital Infections**

Cholestatic pruritus

Chronic graft versus host disease in

liver

Chronic hepatic failure

Chronic hepatitis

Coma hepatic

Cryptogenic cirrhosis

Diabetic hepatopathy

Drug-induced liver injury

Duodenal varices

Focal nodular hyperplasia

Gallbladder varices

Gastric varices

Gastric varices haemorrhage

Graft versus host disease in liver

Haemangioma of liver

Haemorrhagic ascites

Haemorrhagic hepatic cyst

Hepatectomy

Hepatic adenoma

Hepatic atrophy

Hepatic calcification

Hepatic cirrhosis

Hepatic cyst

Hepatic cyst ruptured

Hepatic encelalopathy

Hepatic encephalopathy prophylaxis

Hepatic failure

Hepatic fibrosis

Hepatic fibrosis marker abnormal

Hepatic haemangioma rupture

Hepatic hydrothorax

Hepatic infiltration eosinophilic

Hepatic lesion

Hepatic necrosis

Hepatic steatosis

Hepatitis

Hepatitis acute

Hepatitis cholestatic

Hepatitis chronic active

Hepatitis chronic persistent

Hepatitis fulminant

Hepatitis toxic

Hepatobiliary disease

Hepatocellular foamy cell syndrome

Hepatocellular injury

Hepatopulmonary syndrome

Hepatorenal failure

Hepatorenal syndrome

Hepatotoxicity

Hyperbilirubinaemia

Icterus index increased

Intestinal varices

Ischaemic hepatitis

Jaundice

Jaundice cholestatic

Statistical Analysis Plan 28431754DIA4003

| | | Statistical Final yold Flair 20 13 170 12 11 1003 |
|---|---|---|
| Hepatic Injury | Hypoglycaemia | Male Mycotic Genital Infections |
| Jaundice hepatocellular | | |
| Liver and small intestine transplant | | |
| Liver disorder | | |
| Liver injury | | |
| Lupoid hepatic cirrhosis | | |
| Lupus hepatitis | | |
| Mixed liver injury | | |
| Nodular regenerative hyperplasia | | |
| Non-alcoholic steatohepatitis | | |
| Non-cirrhotic portal hypertension | | |
| Ocular icterus | | |
| Oedema due to hepatic disease | | |
| Oesophageal varices haemorrhage | | |
| Parenteral nutrition associated liver | | |
| disease | | |
| Peripancreatic varices | | |
| Periportal oedema | | |
| Portal hypertension | | |
| Portal hypertensive enteropathy | | |
| Portal hypertensive gastropathy | | |
| Portal triaditis | | |
| Portal vein cavernous transformation | | |
| Portal vein dilatation | | |
| Portopulmonary hypertension | | |
| Radiation hepatitis | | |
| Renal and liver transplant | | |
| Retrograde portal vein flow | | |
| Reye's syndrome | | |
| Reynold's syndrome | | |
| Splenic varices | | |
| Splenic varices haemorrhage | | |
| Subacute hepatic failure | | |
| Varices oesophageal | | |
| Varicose veins of abdominal wall | | |

| Malignancy Bladder Cancer | Malignancy Breast Cancer | Malignancy Phaeochromocytoma |
|---|---|---|
| Bladder adenocarcinoma recurrent | Apocrine breast carcinoma | Phaeochromocytoma |
| Bladder adenocarcinoma stage 0 | Breast angiosarcoma | Phaeochromocytoma crisis |
| - | Breast angiosarcoma | • |
| Bladder adenocarcinoma stage I | metastatic | Phaeochromocytoma excision |
| Bladder adenocarcinoma stage II | Breast cancer | Phaeochromocytoma malignant |
| Bladder adenocarcinoma stage III | Breast cancer female | , |
| Bladder adenocarcinoma stage IV | Breast cancer in situ | |
| Bladder adenocarcinoma stage unspecified | Breast cancer male | |
| Bladder cancer | Breast cancer metastatic | |
| Bladder cancer recurrent | Breast cancer recurrent | |
| Bladder cancer stage 0, with cancer in situ | Breast cancer stage I | |
| Bladder cancer stage 0, without cancer in | _ | |
| situ | Breast cancer stage II | |
| Bladder cancer stage I, with cancer in situ | Breast cancer stage III | |
| Bladder cancer stage I, without cancer in | | |
| situ | Breast cancer stage IV | |
| Bladder cancer stage II | Breast neoplasm | |
| Bladder cancer stage III | Breast sarcoma | |
| Bladder cancer stage IV | Breast sarcoma metastatic | |

| Malignancy Bladder Cancer | <b>Malignancy Breast Cancer</b> | Malignancy Phaeochromocytoma |
|---|---|---|
| Bladder squamous cell carcinoma | | |
| recurrent | Breast sarcoma recurrent | |
| Bladder squamous cell carcinoma stage 0 | Contralateral breast cancer | |
| Bladder squamous cell carcinoma stage I | HER-2 positive breast cancer | |
| | Hormone refractory breast | |
| Bladder squamous cell carcinoma stage II | cancer | |
| | Inflammatory carcinoma of | |
| Bladder squamous cell carcinoma stage III | breast recurrent | |
| | Inflammatory carcinoma of | |
| Bladder squamous cell carcinoma stage IV | breast stage III | |
| Bladder squamous cell carcinoma stage | Inflammatory carcinoma of | |
| unspecified | breast stage IV | |
| unspecifica | Inflammatory carcinoma of | |
| Bladder transitional cell carcinoma | the breast | |
| Bladder transitional cell carcinoma | Intraductal papillary breast | |
| metastatic | neoplasm | |
| Bladder transitional cell carcinoma | Intraductal proliferative breast | |
| recurrent | lesion | |
| Bladder transitional cell carcinoma stage 0 | Invasive breast carcinoma | |
| _ | Invasive ductal breast | |
| Bladder transitional cell carcinoma stage I | carcinoma | |
| | Invasive lobular breast | |
| Bladder transitional cell carcinoma stage II | carcinoma | |
| Bladder transitional cell carcinoma stage | Invasive papillary breast | |
| III | carcinoma | |
| Bladder transitional cell carcinoma stage | Lobular breast carcinoma in | |
| IV | situ | |
| Metastases to bladder | Malignant nipple neoplasm | |
| | Malignant nipple neoplasm | |
| Metastatic carcinoma of the bladder | female | |
| | Malignant nipple neoplasm | |
| Transitional cell carcinoma | male | |
| | Medullary carcinoma of breast | |
| | Metaplastic breast carcinoma | |
| | Metastases to breast | |
| | Mucinous breast carcinoma | |
| | Neuroendocrine breast tumour | |
| | Nipple neoplasm | |
| | Oestrogen receptor positive | |
| | breast cancer | |
| | Paget's disease of nipple | |
| | Phyllodes tumour | |
| | Triple negative breast cancer | |
| | Tubular breast carcinoma | |

| Malignancy Renal Cell Cancer | Malignancy Testicular | Osmotic Diuresis |
|---|---|---|
| Clear cell renal cell carcinoma | Benign neoplasm of testis | Dry mouth |
| Clear cell sarcoma of the kidney | Leydig cell tumour of the testis | Dry throat |
| Denys-Drash syndrome | Sertoli cell testicular tumour | Micturition disorder |
| Hereditary leiomyomatosis renal cell carcinoma | Spermatocytic seminoma | Micturition urgency |
| Hereditary papillary renal carcinoma | Testicle adenoma | Nocturia |
| Metastatic renal cell carcinoma | Testicular cancer metastatic | Pollakiuria |
| Nephroblastoma | Testicular neoplasm | Polydipsia |
| Non-renal cell carcinoma of kidney | Testicular papilloma | Polyuria |
| Renal cancer | Testis cancer | Thirst |
| Renal cancer metastatic | | Tongue dry |
| Renal cancer recurrent | | Urine output increased |
| Renal cancer stage I | | - |
| Renal cancer stage II | | |
| Renal cancer stage III | | |
| Renal cancer stage IV | | |
| Renal cell carcinoma | | |
| Renal cell carcinoma recurrent | | |
| Renal cell carcinoma stage I | | |
| Renal cell carcinoma stage II | | |
| Renal cell carcinoma stage III | | |
| Renal cell carcinoma stage IV | | |
| Rhabdoid tumour of the kidney | | |

| Phimosis | Photosensitivity |
|-------------------|-----------------------------------------------|
| Acquired phimosis | Actinic elastosis |
| Phimosis | Actinic prurigo |
| | Administration site photosensitivity reaction |
| | Application site photosensitivity reaction |
| | Chronic actinic dermatitis |
| | Hartnup disease |
| | Implant site photosensitivity |
| | Infusion site photosensitivity reaction |
| | Injection site photosensitivity reaction |
| | Juvenile spring eruption |
| | Medical device site photosensitivity |
| | Photodermatosis |
| | Photokeratitis |
| | Photoonycholysis |
| | Photosensitivity reaction |
| | Polymorphic light eruption |
| | Solar dermatitis |
| | Solar urticaria |
| | Sunburn |
| | Vaccination site photosensitivity |

| Renal Related | Severe Hypersensitivity/Cutaneous AEs | Upper UTI |
|---|---|---|
| Acute kidney injury | Acute generalised exanthematous pustulosis | Bacterial pyelonephritis |
| | | Emphysematous |
| Acute phosphate nephropathy | Allergic oedema | pyelonephritis |
| Acute prerenal failure | Anaphylactic reaction | Kidney infection |
| Anuria | Anaphylactic shock | Perinephric abscess |
| Azotaemia | Anaphylactic transfusion reaction | Pyelocystitis |
| Blood creatinine increased | Anaphylactoid reaction | Pyelonephritis |
| Blood urea increased | Anaphylactoid shock | Pyelonephritis acute |
| Continuous haemodiafiltration | Angioedema | Pyelonephritis chronic |
| Dialysis | Circulatory collapse | Pyelonephritis fungal |
| Glomerular filtration rate | | |
| decreased | Circumoral oedema | Pyelonephritis mycoplasmal |
| Haemodialysis | Conjunctival oedema | Pyelonephritis viral |
| Haemofiltration | Corneal exfoliation | Pyonephrosis |
| Hypercreatininaemia | Corneal oedema | Renal abscess |
| Neonatal anuria | Cutaneous vasculitis | Renal cyst infection |
| Nephritis | Dermatitis bullous | Urosepsis |
| Nephropathy toxic | Dermatitis exfoliative | |
| Oliguria | Dermatitis exfoliative generalised | |
| Peritoneal dialysis | Drug eruption | |
| Prerenal failure | Drug hypersensitivity | |
| | Drug reaction with eosinophilia and systemic | |
| Renal failure | symptoms | |
| Renal failure acute | Epidermal necrosis | |
| Renal failure neonatal | Epiglottic oedema | |
| Renal impairment | Erythema multiforme | |
| Renal impairment neonatal | Exfoliative rash | |
| | Eye oedema | |
| | Eye swelling | |
| | Eyelid oedema | |
| | Face oedema | |
| | First use syndrome | |
| | Fixed drug eruption | |
| | Gingival oedema | |
| | Gingival swelling | |
| | Gleich's syndrome | |
| | Hereditary angioedema | |
| | Hypersensitivity vasculitis | |
| | Idiopathic angioedema | |
| | Idiopathic urticaria | |
| | Kounis syndrome | |
| | Laryngeal dyspnoea | |
| | Laryngeal oedema | |
| | Laryngospasm | |
| | Laryngotracheal oedema | |
| | Limbal swelling | |
| | Lip exfoliation | |
| | Lip oedema | |
| | Lip swelling Musecutaneous placestion | |
| | Mucocutaneous ulceration | |
| | Mucosa vesicle | |
| | Mucosal erosion | |
| | Mucosal expolicion | |
| | Mucosal releases | |
| | Mucosal ulceration | |
| | Nikolsky's sign | |

| Renal Related | Severe Hypersensitivity/Cutaneous AEs | Upper UTI |
|---------------|---------------------------------------|-----------|
| | Oculomucocutaneous syndrome | |
| | Oculorespiratory syndrome | |
| | Oedema mouth | |
| | Oedema mucosal | |
| | Oral mucosal blistering | |
| | Oral mucosal exfoliation | |
| | Orbital oedema | |
| | Oropharyngeal blistering | |
| | Oropharyngeal swelling | |
| | Palatal oedema | |
| | Penile exfoliation | |
| | Periorbital oedema | |
| | Pharyngeal oedema | |
| | Scleral oedema | |
| | Shock | |
| | Shock symptom | |
| | Skin exfoliation | |
| | Skin necrosis | |
| | Small bowel angioedema | |
| | Stevens-Johnson syndrome | |
| | Stridor | |
| | Swelling face | |
| | Swollen tongue | |
| | Throat tightness | |
| | Tongue exfoliation | |
| | Tongue oedema | |
| | Toxic epidermal necrolysis | |
| | Type I hypersensitivity | |
| | Urticaria | |
| | Urticaria cholinergic | |
| | Urticaria chronic | |
| | Urticaria papular | |
| | Urticarial vasculitis | |
| | Vaginal exfoliation | |

| UTI | Venous Thromboembolic events | Volume Depletion |
|---|---|---|
| Bladder candidiasis | Deep vein thrombosis | Blood pressure decreased |
| Cystitis | Deep vein thrombosis postoperative | Blood pressure orthostatic decreased |
| Cystitis bacterial | Embolism venous | Dehydration |
| Cystitis escherichia | Iliac vein occlusion | Diastolic hypotension |
| Cystitis gonococcal | Inferior vena cava syndrome | Dizziness postural |
| Cystitis haemorrhagic | Inferior vena caval occlusion | Hypotension |
| Cystitis interstitial | Jugular vein occlusion | Hypovolaemia |
| Cystitis klebsiella | Mesenteric vein occlusion | Hypovolaemic shock |
| Cystitis pseudomonal | Obstructive shock | Orthostatic hypotension |
| | Portosplenomesenteric venous | |
| Emphysematous cystitis | thrombosis | Orthostatic intolerance |
| | | Postural orthostatic tachycardia |
| Escherichia urinary tract infection | Post procedural pulmonary embolism | syndrome |
| Fungal cystitis | Postpartum venous thrombosis | Presyncope |
| Funguria | Pulmonary embolism | Shock |
| Genitourinary tract infection | Pulmonary infarction | Shock symptom |
| Streptococcal urinary tract | | |
| infection | Pulmonary microemboli | Syncope |
| Ureter abscess | Pulmonary oil microembolism | Urine output decreased |

Statistical Analysis Plan 28431754DIA4003

| UTI | Venous Thromboembolic events | Volume Depletion |
|---|---|---|
| Ureteritis | Pulmonary thrombosis | |
| Uretheritis | Renal vein embolism | |
| Urethral abscess | Renal vein occlusion | |
| Urethral carbuncle | Subclavian vein thrombosis | |
| Urethral stricture post infection | Vascular occlusion | |
| Urinary bladder abscess | Venous thrombosis | |
| Urinary tract abscess | Venous thrombosis in pregnancy | |
| Urinary tract infection | Venous thrombosis limb | |
| Urinary tract infection bacterial | Visceral venous thrombosis | |
| Urinary tract infection | | |
| enterococcal | | |
| Urinary tract infection fungal | | |
| Urinary tract infection | | |
| pseudomonal | | |
| Urinary tract infection | | |
| staphylococcal | | |

# Appendix 1.4: Adverse Events with Potential Amputation Association

List of selected preferred terms included within the system organ classes of infections and infestations, vascular disorders, nervous system disorders, and skin and subcutaneous tissue disorders

| Infections and Infestations | Vascular Disorders | Nervous System Disorders | Skin and Subcutaneous Tissue<br>Disorders | High Level Term (HLT) Skin and subc | utaneous tissue ulcerations |
|---|---|---|---|---|---|
| Infected skin ulcer | Arteriosclerosis | Paraesthesia | Diabetic ulcer | Penile ulceration | Medical device site erosion |
| Skin infection | Peripheral arterial occlusive disease | Hypoaesthesia | Neuropathic ulcer | Implant site ulcer | Ulcerated haemangioma |
| Staphylococcal skin infection | Peripheral vascular disorder | Diabetic neuropathy | Fungating wound | Cytomegalovirus mucocutaneous ulcer | Incision site erosion |
| Gangrene | Peripheral artery stenosis | Neuropathy peripheral | Diabetic foot | Skin ulcer | Incision site ulcer |
| Osteomyelitis | Peripheral ischaemia | Areflexia | Diabetic neuropathic ulcer | Eyelid erosion | Vaccination site ulcer |
| Diabetic gangrene | Arterial stenosis | Hyporeflexia | Skin erosion | Implant site erosion | Fungating wound |
| Localised infection | Diabetic vascular disorder | Polyneuropathy | | Diabetic foot infection | Ecthyma |
| Wound abscess | Femoral artery occlusion | Autonomic neuropathy | | Application site erosion | Perineal ulceration |
| Wound infection | Thrombosis | Neuropathy peripheral | | Infusion site erosion | Tropical ulcer |
| Subcutaneous abscess | Poor peripheral circulation | Burning sensation | | Mycobacterium ulcerans infection | Injection site erosion |
| Abscess limb | Microangiopathy | Diabetic autonomic neuropathy | | Infusion site ulcer | Pyogenic sterile arthritis<br>pyoderma gangrenosum and acne<br>syndrome |
| Staphylococcal osteomyelitis | Peripheral coldness | Peripheral sensory neuropathy | | Neuropathic ulcer | Scleroderma associated digital ulcer |
| Diabetic foot infection | Diabetic microangiopathy | Peripheral sensorimotor neuropathy | | Skin ulcer haemorrhage | Vulval ulceration |
| Staphylococcal skin infection | Arterial occlusive disease | Sensory disturbance | | Burn infection | Mucocutaneous ulceration |
| Soft tissue infection | Arterial thrombosis | Diabetic neuropathic ulcer | | Diabetic foot | Injection site ulcer |
| Bone abscess | Peripheral artery thrombosis | | | Diabetic ulcer | Pyoderma gangrenosum |
| Osteitis | Arterial occlusive disease | | | Catheter site erosion | Scrotal ulcer |
| Cellulitis | Angiopathy | | | Pyostomatitis vegetans | Application site ulcer |
| Wound <sup>a</sup> | Intermittent claudication | | | Catheter site ulcer | Genital ulceration |
| Dry gangrene | Arterial disorder | | | Medical device site ulcer | Infected skin ulcer |
| Post-operative wound infection | Impaired healing <sup>a</sup> | | | Administration site ulcer | Diabetic neuropathic ulcer |
| Post-operative wound complication <sup>a</sup> | | | | Instillation site erosion | Varicose ulceration |
| Wound dehiscence | | | | Breast ulceration | Vaginal ulceration |
| Burn infection | | | | Instillation site ulcer | Vulvovaginal ulceration |
| Extremity necrosis | | | | Administration site erosion | Auditory meatus external erosion |
| • | | | | Vasculitic ulcer | Skin erosion |
| | | | | Vaccination site erosion | |

<sup>&</sup>lt;sup>a</sup> Although these PTs belong in the SOC of Injury, Poisoning and Procedural Complications or in the SOC of General Disorders and Administration Site Conditions, these terms were retained for the search strategy because of their relevance

# List of preferred terms classified as reversible infections, irreversible infections and osteomyelitis

| Reversible Infections | Irreversible Infections | Osteomyelitis |
|---|---|---|
| Abscess limb | Diabetic gangrene | Bone abscess |
| Burn infection | Dry gangrene | Osteitis |
| Cellulitis | Extremity necrosis | Osteomyelitis |
| Diabetic foot infection | Gangrene | Staphylococcal osteomyelitis |
| Infected skin ulcer | Osteomyelitis | |
| Localised infection | Bone abscess | |
| Skin infection | Osteitis | |
| Soft tissue infection | Osteomyelitis | |
| Staphylococcal skin infection | Staphylococcal osteomyelitis | |
| Subcutaneous abscess | | |
| Wound | | |
| Wound abscess | | |
| Wound dehiscence | | |
| Wound infection | | |